CLINICAL TRIAL: NCT01226381
Title: Comparative Study of the Influence of Two Antagonist Receptors 5-HT3, tropisétron and granisétron, on the Analgesic Effect of Paracétamol
Brief Title: Interaction Between tropisétron / granisétron - paracétamol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0083; 2010-020509-34 (EudraCT Number)
Record Dates: First submitted 2010-10-14; First posted 2010-10-22 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Healthy Volunteers
Keywords: Paracetamol and setrons; No disease, healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Von Frey electronic — This protocol is based on a study of the interaction setron / paracetamol at 4 different levels of plasma concentrations, by repeating the tests at set intervals, while concentrations of setrons down gradually (half-life of 8 to 10 am ) after a single administration. In addition, the interindividual variability of the effects of paracetamol will be studied, and linking with certain genetic polymorphisms reported by the subjects tested

SUMMARY:
This is a Crossover study, double-blind, randomized, controlled versus placebo.

DETAILED DESCRIPTION:
Although the mechanism of action of paracetamol is far from being elucidated, data from the literature suggest that its action would be rather central, without excluding an associated peripheral action. Thus, various studies have shown that paracetamol easily passed the blood-brain barrier. After administration in humans systemically, paracetamol was found in the cerebrospinal fluid.

Various mechanisms have been suggested for the central action. In 1992, Vane and Feirrera have considered the involvement of cyclooxygenase plants, but their conclusions seem to have been invalidated by more recent work showing that, compared to NSAIDs, acetaminophen is a weak inhibitor of these enzymes. Another hypothesized mechanism of action of acetaminophen involves central serotonergic system have demonstrated a reduction of the effect of paracetamol after lesion of descending serotonergic pathways. The inhibition of serotonin synthesis by p-chlorophenylalanine reduced the antinociceptive effect of paracetamol in the hot plate test and formalin test. In addition, paracetamol increases serotonin levels in the cortex and the deck and reduces the number of cortical 5-HT2 receptors, without changing the number of 5-HT1A receptors.

Work done in animals in our laboratory showed a total inhibition of analgesic effects of paracetamol administered orally, intravenously or intrathecally after intrathecal administration of tropisetron, a 5 HT3 receptor antagonist. This suggests a role of 5-HT3 receptor in the mechanism of action of paracetamol, despite the absence of binding of acetaminophen to this receptor.

A clinical trial was conducted in our laboratory in 2004 in 24 healthy volunteers. In this protocol, pain thresholds were measured using a who had been psychophysical test of an electrical nature, the PainMatcher previously validated in our laboratory. This essay has highlighted the pharmacodynamic interaction expected with tropisetron, but also with granisetron.

This difference between the preclinical and clinical results should be studied to determine whether it is due to differences in the mechanism of the analgesic action of paracetamol in humans and animals, or if this is the result administration in clinical doses of granisetron for which it loses its specificity for the 5-HT3 receptor, as in animal studies.

This study is thus complementary to previous work which helped to demonstrate, in humans, the reversion of the analgesic effect of acetaminophen by tropisetron and granisetron.

This protocol is based on a study of the interaction setron -paracetamol at 4 different levels of plasma concentrations, by repeating the tests at set intervals, while concentrations of setrons down gradually (half-life of 8 to 10 am ) after a single administration. In addition, the interindividual variability of the effects of paracetamol will be studied, and linking with certain genetic polymorphisms reported by the subjects tested.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged 18 years and more than 40 years
* Male
* Weight and size within 80 to 120% of theoretical values determined from the Lorentz formula
* Values of vital signs before administering the test products:
* Oral temperature between 35 to 37.5 ° C
* PAS between 100-140 mm Hg
* PAD between 50-90 mm Hg
* Radial pulse between 45-90 beats per minute
* Free from any chronic treatment
* Free of any active disease
* Failure to take any medication within 7 days before enrollment in the study (including no use of analgesics or anti-inflammatory)
* Cooperation and understanding to comply strictly with the requirements of the protocol
* Acceptance to give written consent
* Membership of the scheme of the French Social Security
* Acceptance of registration or the national registry of volunteers participating in research

Exclusion Criteria:

* Contraindications to the administration of paracetamol:
* Known hypersensitivity to paracetamol
* History of hepatitis B or C
* Severe renal insufficiency
* Liver failure
* Contraindications to the administration of tropisetron or granisetron:
* Known hypersensitivity to tropisetron, granisetron, and / or other antagonists of 5-HT3
* Hypertension
* Medical history and / or surgical judged by the investigator or his representative as being incompatible with the test.
* Pathology evolving at the time of assessment for inclusion.
* Excessive consumption of alcohol, tobacco (10 + cigarettes / day), coffee, tea or drinks containing caffeine (equivalent to more than 4 cups per day) or drug addiction.
* Presence of any concurrent treatment (including prescription medicines, vitamins) or taking any medication within 2 weeks before the first administration of the test.
* Topic lacking concentration during workouts nociceptive tests, or presenting training sessions after these tests a low reproducibility of the measured parameters (variability> 20%).
* Topic participating in another clinical trial, or within the period of exclusion or who have received a total compensation of more than 4500 euros for the 12 months preceding the start of the test.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in pain threshold testing mechanical stimulation (von Frey electronic) | Time 0 + 1h, time0 +3h, time 0 +3h30, timet0+12h30, time 0+14h, time0+14h30, time0+23h30, time0+25h, timt0+25h30, time0+34h30, time0+36h, time0+36h30

SECONDARY OUTCOMES:
Assays setrons, paracetamol and its metabolites | Time 0 + 1h, time0 +3h, time 0 +3h30, timet0+12h30, time 0+14h, time0+14h30, time0+23h30, time0+25h, timt0+25h30, time0+34h30, time0+36h, time0+36h30

CONTACTS AND LOCATIONS:
Overall Officials: Claude DUBRAY, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France